CLINICAL TRIAL: NCT00926549
Title: Posterior and Anterior Ocular Imaging With Spectral Domain Optical Coherence Tomography
Brief Title: Ocular Imaging With Spectral Domain Optical Coherence Tomography
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sung Soo Kim, Department of Ophthalmology, Gangnam Severance Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 3-2008-0048
Record Dates: First submitted 2009-05-06; First posted 2009-06-23 (Estimated); Last update posted 2009-06-23 (Estimated); Status verified 2009-06

CONDITIONS: Healthy; Myopia; Hypermetropia
Keywords: spectral domain-OCT; macular thickness; myopia; hypermetropia; normal
MeSH Terms: conditions — Myopia; Hyperopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- spectral domain-OCT (Experimental): Spectral domain-OCT scanning performed.
  Interventions: Device: Spectral domain-OCT (Cirrus™ HD-OCT, Carl Zeiss Meditec AG)

INTERVENTIONS:
Device: Spectral domain-OCT (Cirrus™ HD-OCT, Carl Zeiss Meditec AG) — macular cube scanning
  Other Names: Cirrus™ HD-OCT, Carl Zeiss Meditec AG

SUMMARY:
The purpose of this study is to analyze macular retinal thickness and macular volume using the spectral domain - optical coherence tomography (SD-OCT) in normal eyes and in eyes with various ocular diseases.

DETAILED DESCRIPTION:
Assessment of macular thickness is important for the treatment and follow-up of a variety of ocular diseases. The introduction of optical coherence tomography (OCT) has enabled clinicians to reliably detect small changes in macular thickness and to quantitatively evaluate the efficacy of different therapeutic modalities. In this study using the spectral domain-OCT, we examined the variations of macular retinal thickness and macular volume in normal eyes and in eyes with various ocular diseases.

ELIGIBILITY:
Inclusion Criteria:

* normal eyes
* myopic eyes
* hypermetropic eyes

Exclusion Criteria:

* systemic illness
* cataract
* previous ocular trauma or surgery(other than cataract surgery or refractive surgeries)

Ages: 16 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2009-05; Primary Completion 2009-09 (Estimated); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
macular retinal thickness and volume | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Sung Soo Kim, MD, PhD, Principal Investigator — Department of Ophthalmology, Yonsei University College of Medicine, Gangnam Severance Hospital
Locations (1):
- Yonsei University College of Medicine, Gangnam Severance Hospital, Seoul, South Korea